CLINICAL TRIAL: NCT04174989
Title: MULTI-CENTER,DOUBLE-BLIND, RANDOMIZED, TWO-ARMS, CONTROLLED, PROSPECTIVE CLINICAL INVESTIGATION ASSESSING THE SAFETY AND PERFORMANCE OF A CLASS IIb MEDICAL DEVICE (CLEARPLASMATM) FOR THE TREATMENT OF PATIENTS WITH ACUTE UPPER GASTROINTESTINAL HEMORRHAGE.
Brief Title: Clinical Investigation of Safety and Performance of a Medical Device (ClearPlasma) for the Treatment of Patients With Acute Upper Gastrointestinal Hemorrhage.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PlasFree Ltd. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLAS-01-2019
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Acute Upper Gastrointestinal Hemorrhage; Acute Upper Gastrointestinal Bleeding
Keywords: Acute Upper Gastrointestinal Hemorrhage; Gastrointestinal Hemorrhage; Gastrointestinal Bleeding; Acute Upper Gastrointestinal Bleeding; Plasminogen-Depleted Plasma; Plasma Transfusion
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Intervention Model Description: Multi-center, international, double-blind, randomized, controlled, prospective, first-in-human clinical investigation, in which Patients presenting with acute upper gastrointestinal hemorrhage (AUGIH) and required plasma transfusion, will be randomized to receive a one-time infusion (up to 8 hours) of up to two 250 mL units of PDP (group A) or FFP (group B). The administration of Plasma needs to be in line with the clinical practice and doctor decision.
Who Masked: Participant, Investigator
Masking Description: An unblinded sub-Investigator will prepare the plasma bags to be used for treatment (PDP or FFP). The randomization will be carried out in accordance to the the instructions provided, keeping the Investigator's and Patient's blindness about the content of plasma bags used for transfusion of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasminogen-Depleted Plasma Infusion (Experimental): Patients presenting with acute upper gastrointestinal hemorrhage (AUGIH) and due to undergo a plasma transfusion, will be randomized to receive a one-time infusion (up to 8 hours) of up to two 250 mL units of PDP. In case of transfusions needing more than two units, the third unit and above will consist in regular plasma regardless of treatment group. Patients will be continuously monitored for 8 hours following the transfusion, and will be assessed between 8-12 hours after plasma transfusion or the following morning (the earlier of the two options), between 24-48 hours after plasma transfusion or at discharge (the earlier of the two options) and after 30±3 days after transfusion.
  Interventions: Other: Plasma treated with ClearPlasma (Extra-corporeal plasma filtration device)
- Fresh-Frozen Plasma Infusion (Other): Patients presenting with acute upper gastrointestinal hemorrhage (AUGIH) and due to undergo a plasma transfusion, will be randomized to receive a one-time infusion (up to 8 hours) of up to two 250 mL units of FFP. In case of transfusions needing more than two units, the third unit and above will consist in regular plasma regardless of treatment group. Patients will be continuously monitored for 8 hours following the transfusion, and will be assessed between 8-12 hours after plasma transfusion or the following morning (the earlier of the two options), between 24-48 hours after plasma transfusion or at discharge (the earlier of the two options) and after 30±3 days after transfusion.
  Interventions: Other: Regular fresh-frozen plasma (not treated)

INTERVENTIONS:
Other: Plasma treated with ClearPlasma (Extra-corporeal plasma filtration device) — ClearPlasma is designed to specifically extract plasminogen, a protein that drives fibrinolysis, from up to 250 mL of plasma. ClearPlasma is a non-pyrogenic, sterile, single-use medical device that is indicated for use in conditions where massive bleeding situations exist.
  Arms: Plasminogen-Depleted Plasma Infusion
Other: Regular fresh-frozen plasma (not treated) — Regular fresh-frozen plasma (not treated)
  Arms: Fresh-Frozen Plasma Infusion

SUMMARY:
Pre-market, multi-center, international, double-blind, randomized, controlled, prospective, first-in-human clinical investigation of a Class IIb Investigational Medical Device, in which Patients presenting with acute upper gastrointestinal hemorrhage (AUGIH) and due to undergo a plasma transfusion, will be randomized to receive a one-time infusion (up to 8 hours) of up to two 250 mL units of plasminogen-depleted plasma (PDP) or fresh-frozen plasma (FFP).

In case of transfusions needing more than two units, the third unit and above will consist in regular plasma for both treatment groups. Patients will be continuously monitored for 8 hours following the transfusion, and will be assessed between 8-12 hours after plasma transfusion or the following morning (the earlier of the two options), between 24-48 hours after plasma transfusion or at discharge (the earlier of the two options) and after 30+/-3 days after transfusion.

DETAILED DESCRIPTION:
Upper gastrointestinal hemorrhage (UGIH) is one of the most common gastrointestinal emergencies, and is associated with significant morbidity and mortality. Acute upper gastrointestinal hemorrhage (AUGIH) management guidelines call for aggressive hemodynamic resuscitation, prevention and treatment of complications and treatment of bleeding, which generally includes endoscopic intervention and transfusion of appropriate blood components. However, in many cases, spontaneous hyperfibrinolysis occurs, jeopardizing pharmacological control of AUGIH. Antifibrinolytic drugs are considered effective in counteracting hyperfibrinolysis, but are associated with various side effects, such as neurotoxicity and accelerated fibrinolysis upon prolonged use.

Fibrin clot breakdown is actively mediated by plasmin, a serine protease which cleaves fibrin. Administration of plasma depleted of plasminogen, the precursor of plasmin, may shift the balance towards coagulation.

PlasFree Ltd. has developed ClearPlasma, a single-use, extracorporeal plasma filtration device which extracts plasminogen from plasma to reduce fibrinolysis. The resulting plasminogen-depleted plasma (PDP) is expected to reduce risk of fibrinolysis and re-bleeding in Patients undergoing plasma transfusions.

The Primary Objective of this trial is to assess the safety profile of a one-time infusion of up to two units of PDP obtained through filtration with ClearPlasma in Patients presenting with acute upper gastrointestinal hemorrhage and to compare it to the same procedure carried out using FFP units.

The Secondary Objective of this trial is to assess the efficacy of a one-time infusion of up to two units of PDP obtained through filtration with ClearPlasma in the reduction of re-bleeding in Patients presenting with acute upper gastrointestinal hemorrhage (as a measure of the performance of ClearPlasma) and to compare it to the same procedure carried out using FFP units.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Patients.
2. Patients aged ≥ 18 and ≤ 80 years old.
3. Patients presenting with acute upper gastrointestinal hemorrhage (> 0.5 L), diagnosed by presence of blood in gastric lavage, hematemesis or melena within no longer than 24 h before enrolment.
4. Patients presenting with acute upper gastrointestinal hemorrhage (< 24 h) for which fresh frozen plasma (FFP) has been ordered.
5. Patients understanding the nature of the study and providing their informed consent to participation.
6. Patients willing and able to attend the follow-up visits and procedures foreseen by study protocol.

Exclusion Criteria:

1. Patients who underwent a plasma infusion in the 30 days before enrolment.
2. Patients in a life-threatening condition at the time of enrolment.
3. Patient on anticoagulant therapy at the time of enrolment.
4. Patients with known renal failure (creatinine clearance < 30 mL/min) at the time of enrolment.
5. Patients suffering of Hemophilia A or B.
6. Patients suffering of venous and arterial thromboembolic events within 3 months before the enrolment.
7. Patients with history of allergic reaction to plasma, polyethersyplone or polycarbonate.
8. Patients suffering of IgA deficiency at the time of enrolment.
9. Patients with history of hemorrhage while on anticoagulant treatment (warfarin, apixaban, rivaroxaban, dabigatran, low molecular weight heparin).
10. Patients identified by the Investigator to have any underlying medical conditions that may preclude conduct of study procedure (i.e. making the administration of study treatment hazardous) or obscure the interpretation of safety objectives.
11. Patients who are participating or have participated in other clinical studies within the 30 days before the study enrolment.
12. Women who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical investigation and for 3 months later.
13. Female Patients of childbearing age (less than 24 months after the last menstrual cycle) who do not use adequate contraception *.

    * Methods at low risk of contraceptive failure (less than 1% per year) when used consistently, including: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), some intra-uterine devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-10-24 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-13 (Actual)

PRIMARY OUTCOMES:
Safety Profile in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient).
  Comparison of adverse events rate during the study period and within 30±3 days after transfusion with PDP (group A) or FFP (group B). All adverse occurrences (serious/non-serious or device-related/non-device related) will be recorded prospectively, categorized and evaluated for causality using defined criteria.

SECONDARY OUTCOMES:
Incidence of re-bleeding episodes in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient).
  Comparison of the number of re-bleeding episodes occurring for the Patient throughout the study period and within 30±3 days after transfusion with PDP (group A) or FFP (group B).
Duration of hospital stay in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient) or until patient discharge.
  Comparison of the duration of the hospital stay for the Patient up to 30±3 days after transfusion with PDP (group A) or FFP (group B).
CBC profile in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient).
  Comparison of complete blood count (CBC) profiles between Patients who received transfusion with PDP (group A) or FFP (group B) at baseline (Screening Visit) versus T=8-12h, T=24-48h and End of Study Visit.
D-dimer profile in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient).
  Comparison of D-dimer profiles between Patients who received transfusion with PDP (group A) or FFP (group B) at baseline (Screening Visit) versus T=8-12h, T=24-48h and End of Study Visit.
PT/INR (blood coagulation parameter) measurement in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient) or until patient discharge.
  Comparison of Prothrombin Time and International Normalized Ratio (PT/INR) between Patients who received transfusion with PDP (group A) or FFP (group B) until Patient discharge from hospital.
aPTT (blood coagulation parameter) measurement in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient) or until patient discharge.
  Comparison of Activated Partial Thromboplastin Time (aPTT) between Patients who received transfusion with PDP (group A) or FFP (group B) until Patient discharge from hospital.
Incidence of venous and arterial thromboembolic events in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient).
  Comparison of the incidence of venous and arterial thromboembolic events during the study period and within 30±3 days after transfusion with PDP (group A) or FFP (group B).
Plasma transfusion-related mortality in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient).
  Comparison of the plasma transfusion-related mortality during the study period and within 30±3 days after transfusion with PDP (group A) or FFP (group B).
Total blood loss from transfusion in Patients treated with PDP versus FFP. | Entire Study Period (up to 1 month per patient) or until patient discharge.
  Comparison of total blood loss from transfusion with PDP (group A) or FFP (group B) until Patient discharge from hospital, as measured by:
  1. Red blood cells (RBC) units transfused;
  2. Plasma units transfused;
  3. Platelet units transfused;
  4. Hemoglobin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Franceschi, MD, Principal Investigator — Chief of Emergency Medicine Fondazione Policlinico Universitario A. Gemelli IRCCS Università Cattolica del Sacro Cuore Largo A. Gemelli
Locations (8):
- Czechia (3):
  - Charles University Teaching Hospital, Hradec Králové
  - University Hospital in Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
- Israel (3):
  - Wolfson Medical center, Holon
  - Department of Surgery B, Meir Medical Center Kfar Saba, Kfar Saba
  - Department of Surgery, Rabin Medical Center, Petah Tikva
- Italy (2):
  - S.C. di Anestesia e Rianimazione 1, Azienda Ospedaliera Universitaria Policlinico di Modena, Modena
  - Area Medicina D'Urgenza e Pronto Soccorso, Fondazione Policlinico Universitario A. Gemelli, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arya RC, Wander G, Gupta P. Blood component therapy: Which, when and how much. J Anaesthesiol Clin Pharmacol. 2011 Apr;27(2):278-84. doi: 10.4103/0970-9185.81849. PMID 21772701
- [Background] Demarmels Biasiutti F, Sulzer I, Stucki B, Wuillemin WA, Furlan M, Lammle B. Is plasminogen deficiency a thrombotic risk factor? A study on 23 thrombophilic patients and their family members. Thromb Haemost. 1998 Jul;80(1):167-70. PMID 9684804
- [Background] Hirayama F. Current understanding of allergic transfusion reactions: incidence, pathogenesis, laboratory tests, prevention and treatment. Br J Haematol. 2013 Feb;160(4):434-44. doi: 10.1111/bjh.12150. Epub 2012 Dec 6. PMID 23215650
- [Background] Matei D, Groza I, Furnea B, Puie L, Levi C, Chiru A, Cruciat C, Mester G, Vesa SC, Tantau M. Predictors of variceal or nonvariceal source of upper gastrointestinal bleeding. An etiology predictive score established and validated in a tertiary referral center. J Gastrointestin Liver Dis. 2013 Dec;22(4):379-84. PMID 24369318
- [Background] Pandey S, Vyas GN. Adverse effects of plasma transfusion. Transfusion. 2012 May;52 Suppl 1(Suppl 1):65S-79S. doi: 10.1111/j.1537-2995.2012.03663.x. PMID 22578374
- [Background] Rockall TA, Logan RF, Devlin HB, Northfield TC. Incidence of and mortality from acute upper gastrointestinal haemorrhage in the United Kingdom. Steering Committee and members of the National Audit of Acute Upper Gastrointestinal Haemorrhage. BMJ. 1995 Jul 22;311(6999):222-6. doi: 10.1136/bmj.311.6999.222. PMID 7627034
- [Background] Rubinstein LV, Steinberg SM, Kummar S, Kinders R, Parchment RE, Murgo AJ, Tomaszewski JE, Doroshow JH. The statistics of phase 0 trials. Stat Med. 2010 May 10;29(10):1072-6. doi: 10.1002/sim.3840. PMID 20419759
- [Background] Schuster V, Hugle B, Tefs K. Plasminogen deficiency. J Thromb Haemost. 2007 Dec;5(12):2315-22. doi: 10.1111/j.1538-7836.2007.02776.x. Epub 2007 Sep 26. PMID 17900274
- [Background] Association of Anaesthetists of Great Britain and Ireland; Thomas D, Wee M, Clyburn P, Walker I, Brohi K, Collins P, Doughty H, Isaac J, Mahoney PM, Shewry L. Blood transfusion and the anaesthetist: management of massive haemorrhage. Anaesthesia. 2010 Nov;65(11):1153-61. doi: 10.1111/j.1365-2044.2010.06538.x. PMID 20963925
- [Background] Wilkins T, Khan N, Nabh A, Schade RR. Diagnosis and management of upper gastrointestinal bleeding. Am Fam Physician. 2012 Mar 1;85(5):469-76. PMID 22534226
- See also: PlasFree Ltd. official website — https://www.plas-free.com/